CLINICAL TRIAL: NCT00251160
Title: Arthroscopic Electrothermal Capsulorrhaphy, ETAC, Versus Open Inferior Capsular Shift, ICS in Patients With Shoulder Instability: A Multicentre Randomized Clinical Trial
Brief Title: Electrothermal Arthroscopic Capsulorrhaphy (ETAC) and Open Inferior Capsular Shift in Patients With Shoulder Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Arthritis Society, Canada (Other); Smith and Nephew (formerly Oratec Interventions) (Unknown)
Responsible Party: Principal Investigator, Dr. Nicholas Mohtadi, Clinical Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10650; MCT-64671 (CIHR) (Other Grant/Funding Number: Canadian Institutes of Health Research); ISRCTN68224911 (Registry Identifier: Current Controlled Trials)
Record Dates: First submitted 2005-11-07; First posted 2005-11-09 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Shoulder Dislocation
Keywords: Multi-directional instability; MDI; Ligamentous laxity; Multi-directional laxity; MDL-AII; Shoulder instability; electrothermal capsulorrhaphy, ETAC; inferior capsular shift, ICS; capsular redundancy
MeSH Terms: conditions — Shoulder Dislocation; Joint Instability

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ETAC (Active Comparator)
  Interventions: Procedure: Electrothermal arthroscopic capsulorrhaphy (ETAC)
- Open ICS (Active Comparator)
  Interventions: Procedure: Open inferior capsular shift (ICS)

INTERVENTIONS:
Procedure: Electrothermal arthroscopic capsulorrhaphy (ETAC) — The Oratec Vulcan Generator electro-thermal system (Oratec Interventions Inc., Menlo Park, CA, USA) delivers heat at 75C and 40 watts. An anterior portal is established above the superior border of the subscapularis tendon. For MDI patients, the heat probe is introduced through the posterior portal. The capsule is shrunk using a grid pattern until excess volume is diminished. The extent of the heat probe application is identical to the landmarks used for the open ICS. Care is taken to avoid applying heat to the capsule in the region from 5-7 o'clock within 1cm of the glenoid rim to avoid the axillary nerve. The method of heat application utilizes a grid pattern, which is less likely to cause dissolution of the capsule and subsequent catastrophic capsular loss.
  Other Names: Heat probe
  Arms: ETAC
Procedure: Open inferior capsular shift (ICS) — MDI: lateral capsule released antero-superiorly from rotator interval to equator, posteriorly on the humeral neck. MDL-AII: release from the rotator interval to 7 o'clock (Right) or 5 o'clock (Left) position on humeral neck, to tighten the 2 bands of the inferior GH ligaments, middle GH ligament and rotator interval. Bone adjacent to the articular surface on the surgical neck of the humerus is roughened to create a bleeding bony bed. With the arm in 0deg flexion, 30deg abduction, 30deg external rotation, the inferior leaflet of the capsule is shifted superiorly and slightly laterally, and sutured to the rim of the capsule using a non-absorbable suture. Superior leaflet is shifted inferiorly and sutured. Subscapularis is repaired at its anatomic length using interrupted sutures.
  Other Names: Open inferior capsular shift
  Arms: Open ICS

SUMMARY:
This trial will compare the effectiveness of electrothermal arthroscopic capsulorrhaphy (ETAC) to the current reference standard procedure, open inferior capsular shift (ICS), for the treatment of shoulder instability caused by ligamentous capsular redundancy. Multi-directional instability (MDI) and multi-directional laxity with anteroinferior instability (MDL-AII) are the two types of shoulder instabilities included in this trial.

Hypothesis: There is no difference in disease-specific quality of life between patients undergoing an ETAC versus an open ICS for the treatment of shoulder instability caused by capsular ligamentous redundancy.

DETAILED DESCRIPTION:
The shoulder is the most frequently dislocated joint in the body. Multiple causes and pathologies account for the various types of shoulder instability. Multi-directional instability (MDI) and multi-directional laxity with anteroinferior instability (MDL-AII) are similar in pathology, less common and more difficult to treat. These types of shoulder instability are caused by ligamentous capsular redundancy. When non-operative management fails for these patients, their quality of life is significantly impaired and surgical treatment is required to tighten the loose ligaments and joint capsule. A new way to treat these patients involves arthroscopic thermal shrinkage of the tissue to tighten the joint. However, there is a lack of scientific evidence to support the use of this technique called, electrothermal arthroscopic capsulorrhaphy (ETAC). The current reference (gold) standard treatment for these patients is an open inferior capsular shift (ICS) procedure. Therefore, this trial will compare the effectiveness of these surgical techniques (ETAC vs. ICS) in patients with MDI and MDL-AII by determining patient related quality of life.

This study is designed as a multicentre, randomized controlled trial. Patients diagnosed with either MDI or MDL-AII who failed standardized non-operative management will undergo a diagnostic shoulder arthroscopy, and if appropriate, will be subsequently randomized in the operating room to either an ETAC or ICS surgical procedure. Computer-generated, stratified block randomization is used. Stratification is based on two variables:

1. surgeon - to account for any differences between surgeons, and
2. diagnosis (MDI or MDL-AII) - to account for any differences in the severity of pathology.

The disease-specific quality of life is assessed using a validated questionnaire, the Western Ontario Shoulder Instability Index, measured at baseline, and 3, 6, 12 and 24 months. The WOSI index has 21 questions, divided into four categories to assess physical symptoms, sport/recreation/work, lifestyle and emotions. Each question is scored out of 100 using a visual analog scale response format. A lower score reflects a better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Ages 14 years or greater
* Diagnosis of MDI or MDL-AII. Diagnosis will require two or more of the following:

  * Symptomatic translation (pain or discomfort) in one or more directions: anterior, inferior and/or posterior;
  * Ability to elicit unwanted glenohumeral translations that reliably produce symptoms with one of the following tests: the anterior and posterior apprehension tests, the anterior and posterior load and shift tests, the fulcrum test, the relocation test, the Fukuda test, and/or the push-pull or stress test with the patient supine;
  * Presence of a positive sulcus sign of 1 centimetre or greater gap that reproduces the patient's clinical symptoms of instability and should be both palpable and visible;
  * Symptoms of instability: subluxation or dislocation.
* Written informed consent
* Failed at least 6 months of non-operative treatment
* Confirmed capsular-ligamentous redundancy as determined by diagnostic arthroscopy examination.

Exclusion Criteria:

* Neurologic disorder (ie: axillary nerve injury; syringomyelia)
* Cases involving third party compensation
* Patients with primary posterior instability
* A bony abnormality (Hill Sachs/bony Bankart) on standard series of x-rays consisting of a minimum of an anteroposterior view, lateral in the scapular plane and an axillary view
* Presence of a Bankart lesion on arthroscopic exam of the joint
* Presence of an unstable biceps anchor (ie: superior labral anterior and posterior [SLAP] lesion) on arthroscopic exam of the joint
* Presence of a full-thickness rotator cuff tear.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 1999-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Western Ontario Shoulder Instability (WOSI) Index | Baseline, 3, 6, 12, 24 months post-operatively

SECONDARY OUTCOMES:
Constant score (European Shoulder Society) | Baseline, 3, 6, 12, 24 months post-operatively
Recurrent instability | Up to 24 months post-operatively
Complications | Intra-operatively and up to 8 weeks post-operatively
Operative time | Day of surgery
American Shoulder and Elbow Surgeon's Score (ASES) | Baseline, 3, 6, 12, 24 months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Mohtadi, MD, FRCSC, Principal Investigator — University of Calgary Sport Medicine Centre
Locations (7):
- Canada (7):
  - University of Calgary Sport Medicine Centre, Calgary, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Pan Am Medical and Surgical Centre, Winnipeg, Manitoba
  - Hamilton General Hospital, Hamilton, Ontario
  - Fowler Kennedy Sport Medicine Centre, London, Ontario
  - St. Joseph's Health Centre, London, Ontario

REFERENCES:
- [Background] Mohtadi NG, Hollinshead RM, Ceponis PJ, Chan DS, Fick GH. A multi-centre randomized controlled trial comparing electrothermal arthroscopic capsulorrhaphy versus open inferior capsular shift for patients with shoulder instability: protocol implementation and interim performance: lessons learned from conducting a multi-centre RCT [ISRCTN68224911; NCT00251160]. Trials. 2006 Feb 2;7:4. doi: 10.1186/1745-6215-7-4. PMID 16542033
- [Result] Mohtadi NG, Kirkley A, Hollinshead RM, McCormack R, MacDonald PB, Chan DS, Sasyniuk TM, Fick GH, Paolucci EO; Joint Orthopaedic Initiative for National Trials of the Shoulder-Canada. Electrothermal arthroscopic capsulorrhaphy: old technology, new evidence. A multicenter randomized clinical trial. J Shoulder Elbow Surg. 2014 Aug;23(8):1171-80. doi: 10.1016/j.jse.2014.02.022. Epub 2014 Jun 15. PMID 24939380
- See also: Study protocol and Lessons learned from conducting a multi-centre RCT, in online journal "Trials" — http://www.trialsjournal.com/content/7/1/4